CLINICAL TRIAL: NCT00737620
Title: Evaluation of Heparin Bonded Vascular Graft Versus Standard Graft in Prosthetic Arteriovenous Access for Hemodialysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Dr David Shemesh, Dr, Shaare Zedek Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11111
Record Dates: First submitted 2008-08-17; First posted 2008-08-19 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2011-12

CONDITIONS: Hemodialysis Fistula Thrombosis
Keywords: Renal Failure, End Stage; Blood Vessel Grafting; Hemodialysis; Surgical Arteriovenous Shunt
MeSH Terms: conditions — Kidney Failure, Chronic; Arteriovenous Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- propaten graft (Active Comparator)
  Interventions: Procedure: Prosthetic AV graft implantation
- Standard graft (Active Comparator)
  Interventions: Procedure: Prosthetic AV graft implantation

INTERVENTIONS:
Procedure: Prosthetic AV graft implantation — Surgical arteriovenous fistula creation with standard or propaten graft

SUMMARY:
The majority of bridge graft fistula with polytetrafluoroethylene (PTFE) for hemodialysis access will develop stenosis at the venous anastomosis and eventually will fail. Aspirin have been used for many years as a prophylactic drug therapy to prevent thrombosis but good clinical evidence for its benefit is lacking. Many drugs have been used to reduce intimal hyperplasia in animal models. Until recently there has been little success in clinical trials of anti-inflammatory, antiproliferative, antiplatelet, antithrombotic or calcium channel blocking drugs. Recently a major breakthrough was done by GORE when introducing the new heparin bonded PTFE graft by covalent attachment. This trial is planed to assess and compare between the GORE-TEX® PROPATEN vascular graft versus unmodified ePTFE grafts the patency and complication.

ELIGIBILITY:
Inclusion Criteria:

* All the patients who are scheduled for the creation of a new prosthetic access with informed consent will be enrolled in the trial
* Investigators will attempt to enroll a male:female ratio of patients representative of their current patient population

Exclusion Criteria:

* Anticoagulation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2008-03; Primary Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Patency of AV fistula | Study period

CONTACTS AND LOCATIONS:
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Jerusalem, Israel

REFERENCES:
- [Derived] Shemesh D, Goldin I, Hijazi J, Zaghal I, Berelowitz D, Verstandig A, Olsha O. A prospective randomized study of heparin-bonded graft (Propaten) versus standard graft in prosthetic arteriovenous access. J Vasc Surg. 2015 Jul;62(1):115-22. doi: 10.1016/j.jvs.2015.01.056. Epub 2015 Mar 12. PMID 25770987